CLINICAL TRIAL: NCT05498454
Title: Differential Contributions of Online Stress and Pain-explicit Mindfulness Treatment Groups to Processes, Patient Experience and Outcomes in Chronic Pain: A Randomized Controlled Trial and Qualitative Analysis
Brief Title: Contribution of Online Stress and Pain Mindfulness Treatment to ACT Process Change and Outcomes in Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Government of Jersey (Other Government)
Collaborators: Liverpool John Moores University (Other); Breathworks CIC (Unknown); Primary Care Body (Jersey, United Kingdom) (Unknown)
Responsible Party: Principal Investigator, Dr Alessio Agostinis, Consultant Clinical Psychologist, Government of Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MT/LC 11/10/2019
Record Dates: First submitted 2022-07-21; First posted 2022-08-12 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain
Keywords: mindfulness; chronic pain; pain; Acceptance and Commitment Therapy
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Health

STUDY DESIGN:
Intervention Model Description: waiting list controlled - then waiting list randomly allocated to one or two possible treatments. Effectively, one Arm, then splitting into two ( 1 + 2)
Who Masked: Outcomes Assessor
Masking Description: The data analysis will be performed blind by one of the researchers - after data has been anonymised and transferred.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breathworks Mindfulness for Health (Active Comparator): an 8-week, online, protocol based mindfulness course designed to manage chronic pain and chronic health conditions
  Interventions: Behavioral: Breathworks Mindfulness (Health or Stress Arm)
- Breathworks Mindfulness for Stress (Active Comparator): an 8-week, online, protocol based mindfulness course designed to manage stress
  Interventions: Behavioral: Breathworks Mindfulness (Health or Stress Arm)
- Waiting list (No Intervention): The Waiting list will be for the whole sample of participants (acting as a waiting list control). From this, participants will be randomly allocated to one of the Arms above

INTERVENTIONS:
Behavioral: Breathworks Mindfulness (Health or Stress Arm) — As for previous descriptions
  Arms: Breathworks Mindfulness for Health; Breathworks Mindfulness for Stress

SUMMARY:
Mindfulness is a popular set of knowledge and practical techniques that can help people cope with stress. It includes meditation practices, everyday small practices to break and change usual habits, as well as understanding and developing competencies to be more aware of thoughts, emotions and physical sensations. Mindfulness can help not to excessively react to them, or becoming distressed by these, as well as pain.

In persistent pain (pain that lasts more than three months), mindfulness is thought to improve depression, quality of life, and even how sore people feel.

There are numerous versions of mindfulness and mindfulness-based therapies. One approach, Acceptance and Commitment Therapy (ACT), is based on science (as opposed to religion or common sense). ACT helps people to learn about and apply skills to cope with thoughts, emotions and sensations without getting upset, distracted or impeded by them. It also assists people to develop the ability to set clear goals that matter in their life. ACT evaluates successful outcomes in this areas (called 'processes') and how these link to changes in pain, mood and stress. However, more puritan mindfulness courses tend to only focus on the latter.

Research on mindfulness courses for chronic pain, can show that people improve, but not so well what changes in people's experience and skills, or how such skills are applied. The investigators also know that pain sufferers who attend mindfulness courses for stress, may say it is not so relevant to their pain difficulties.

In this study the investigators want to explore how both mindfulness for stress and mindfulness for pain courses, online, contribute to:

* How specific areas of ACT and other mindfulness learning change
* If/how these link with practical skills and any emotional or improvements in the participants' quality of life, use of medication or GP visits.
* If/how the above correlate with physiological stress responses such a heart rate variability To help us evaluate this, the investigators will ask participants to complete scientifically accepted questionnaires and interview a proportion of participants. Some may be invited to wear portable heart rate monitors. The investigators will then use statistical methods and qualitative methods to evaluate change.

This may help us with better supporting chronic pain sufferers with choices around mindfulness as a standalone or as part of attending intensive pain-coping programmes involving different professions.

DETAILED DESCRIPTION:
Detailed Description

Mindfulness can be defined operationally as Paying attention; on purpose in the present moment and non-judgmentally.

Evidence-based (often referred to as 'secular') mindfulness has seen an exponentially increasing interest in the scientific literature and the estimated number of published scientific journals has recently been reported to have grown from one single journal in 1982, to 667 scientific publications in 2016 and in excess of 30,000 Media Pieces in Newspapers.

However, there are unknowns around the mechanisms (the 'vehicles' of change) by which mindfulness works. These must be better understood in order to avoid continued professional and public misinformation, poor research and ultimately, potential harm to the end user. (Van Dam, van Vugt et al. 2018).

ISSUES WITH AND IMPLICATIONS OF WHAT THE INVESTIGATORS CURRENTLY DEFINE AS MINDFULNESS AND ITS APPLICATION TO CHRONIC PAIN

Within the context of the exponential growth of interest in and research of mindfulness including in the treatment of chronic pain, several factors have contributed to the consideration for the current project:

1. The integration of mindfulness based interventions in gold-standard multidisciplinary treatments for chronic pain, such as ACT.
2. Researchers' calls to improve intention to treat, to better understand facets of what is understood to be mindfulness, better targetting of and a more unified approach to mindfulness-change process variables - thus aiming to reduce treatment burden.
3. There are relevant mindful mechanisms and processes specifically in chronic pain that have made a case from both the ACT and the more purist mindfulness research derived from group based interventions or meditation alone in chronic pain - and that are not currently typically or routinely included in mindfulness groups research for chronic pain.
4. Methodological issues including

   1. lack of clarity about providers' competencies and requirements in chronic pain,
   2. arbitrary removal of essential components of a given intervention,
   3. often no active or waiting list control condition and
   4. no consideration at all of utilising a theoretically valid and coherent process-measurement frameworks nor consideration for the teachers' competencies requirements when delivering mindfulness courses to chronic pain patients

      From reviewing the evidence quoted, the research on mindfulness for chronic pain has exclusively utilised standardised mindfulness groups typically aimed at stress populations, excluded less researched pain explicit (contextually relevant to pain) mindfulness group interventions, ignored theoretically valid mindful-process measurement provided by frameworks such as the ACT framework, or not controlled appropriately for significant confounding factors.

      This debate is increasingly important considering that recently published audit data suggests that mindfulness in one format or the other, or as part of ACT-based multidisciplinary treatment is being provided regularly in pain management centres in the UK . This has been leading, possibly prematurely, to discussion about providing training in mindfulness competencies for pain practitioners such as mindfulness enquiry or leading meditations, which may lead, in turn, to implementing professional skills without sound, targeted and theoretically evidenced rationale.

      METHODOLOGICAL ISSUES WITH CURRENT MINDFULNESS RESEARCH AND THE IMPROVEMENTS WITH THIS STUDY

      The current research will therefore aim to address and control, some of the currently reported methodological issues in research on group mindfulness based interventions (MBIs), including:
      * Utilising a waiting list for the whole group as a control prior to randomisation. This will act as a pseudo treatment-as-usual condition and will track key outcome and process measures across this time.
      * Utilising two active interventions, Mindfulness for Stress (MfS) and Mindfulness for Health-Mindfulness Based Pain Management (MfH-MBPM), with a standardised, transparent, comparable in content, time and delivery process that can therefore be easily evaluated for adherence and treatment fidelity.
      * Using established and matched teacher's competence in line with UK Network standards for the intervention delivered.
      * Utilising the same 'dosage' and type of interventions (groups with similar structure, delivery times and requirements for practice) utilising MfH-MBPM and MfS protocols, teacher notes and processes that are standardised
      * Inter-rater reliability assessment of fidelity to the treatment provided
      * Using appropriate psychometric and qualitative analysis and targeting of explicit process-change.
      * Reporting adverse side effects
      * Measures in line with IMMPACT recommendations for research on chronic pain
      * the investigators may also submit Ethics amendments to include Heart Variability Measurement in a proportion of the study cohort, to have a biological correlate.

      Identified Risks Likelihood Potential Impact/Outcome Risk Management/Mitigating Factors:

      Practicing mindfulness meditation has been known to trigger distressing memories in patients with existing Trauma/PTSD

      Low

      Participant:

      • Psychological Stress

      Researcher
      * Anxiety about dealing with a complex situation • Exclusion criteria for enrolling in the study will include those with pre-existing psychiatric comorbidities, particularly Trauma/PTSD conditions
      * As the investigators are recruiting from primary care GPs will be informed of this criteria as will patients themselves in their information packs
      * The researcher will be able to signpost participant to the relevant support services

      Discussion of sensitive topics in interview has potential to cause distress to participant

      Low Participant:

      • Psychological Stress

      Researcher
      * Anxiety about dealing with a complex situation • Offer to cease interview
      * Exclusion criteria (as above)
      * The researcher will be able to signpost participant to the relevant support services

      Conflict between participants in group setting

      Low Participant:

      • Psychological Stress

      Researcher
      * Anxiety about dealing with a complex situation
      * The researcher will have the necessary training and experience in group facilitation to handle conflicts

      Data collection & interviews may possibly take place in an unfamiliar location with people not already known to the researcher

      High

      Researcher
      * Physical Injury or Psychological Harm • Visit location prior to data collection to assess possible risks associated with built and social environment
      * Use this information to plan session
      * Identify back up at location or online preferably
      * Allow extra time to familiarise participants with research and environment
      * Researcher to have contact details and means of making timely contact with back up

      Disclosure of information about poor practice

      Low Immediate, urgent or prompt response may be required from service providers • Ensure all verbal and written information about research indicates possible researcher response to disclosure

      • The researcher will be able to signpost participant to the relevant support services

      Disclosure of unmet health or social care needs

      Medium Immediate, urgent or prompt response may be required from service providers • Ensure all verbal and written information about research indicates possible researcher response to disclosure

      • The researcher will be able to signpost participant to the relevant support services

      Research participant in danger of harm to self or others

      Low Immediate, urgent or prompt response may be required from service providers • Ensure all verbal and written information about research indicates possible researcher response to disclosure

      • The researcher will be able to signpost participant to the relevant support services

      STATISTICAL POWER This study will be a modification of a previous pilot test trial of a brief, widely inclusive UK primary care setting (McCracken, Sato and Taylor, 2013), to include the whole sample of participants acting as a waiting list control, randomly allocated to two active treatment conditions. In line with this study which was delivered in a population area of 119,000 people, power calculations were not completed, nor were formal predictions of significant treatment effects. This was on the basis that the same treatment format and in a community based sample had not been tried before and demonstrated of successful recruitment of > 60 participants within a two-month period and reporting moderate effect sizes for the active condition. Given the whole island population of Jersey (N.B. this is United Kingdom Jersey - not US) is estimated currently at 106,000, power calculations will not be provided in this study as the sample size was deemed appropriate in the previous that also cited a number of studies with similar sample sizes and obtained from populations greater than Jersey.

      Plan for missing data to address situations where variables are reported as missing, unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results: The investigators will utilise mean substitution for missing items or alternative substitution technique.

      The quantitative analysis will be also bolstered by a qualitative study:

      DESIGN AND SETTING A qualitative study involving semi-structured interviews will be held, with a topic guide informed by the ACT psychological flexibility model and Day's framework for mindfulness-relevant processes in chronic pain, and based on mindfulness research improvement based on adaptations of Mindfulness Based Cognitive Therapy (MBCT) for chronic pain

      Exclusion criteria (in addition to quantitative study criteria):

      Non-completers (participants who completed less than 6/8 course sessions) Declined to take part in interviews

      SAMPLING An opportunity sample from all patients invited to take part to the quantitative research aspect, invited as part of the initial quantitative study informed consent process.

      We will invite all participants from the sample, aiming from 10-15 participants from each the stress and pain version of the courses, hence a total sample of 30 participants maximum and a target of 10 completed interviews for each intervention.

      N.B. This study's initial Ethics Submission was for a face to face project in February 2019. However, due to Covid-19 and lack of funding, the investigators requested and agreed Ethics amendments to go online. These amendments were approved by the Jersey Healthcare Ethics Committee after submission on 24/05/2022, their meeting on 26/05/2022 and formal email of approval on 30/05/2022.

ELIGIBILITY:
Once potential participants have consented, searches will be run on GP electronic health records to identify suitability. Demographic data including gender, age, ethnicity and employment status, pain diagnoses, current medication and dosage, co-morbidities and mental health diagnoses will be extracted via GP referral to the study, including that the patients meet inclusion criteria and do not meet any of the exclusions.

INCLUSION CRITERIA

* Diagnosis of Chronic Pain: Pain for longer than 3 months
* Ability to communicate and literacy in English
* Age 18 years or older
* No current outstanding medical tests or procedures for conditions expected by the GP to interfere with participation in treatment.
* Has not previously received non-medical treatment at a specialist pain centre, or attended a multidisciplinary pain management programme.
* Ability to utilise online video conferencing technology (i.e. ownership of a compatible device & necessary technical competence)

EXCLUSION CRITERIA

* Patients who are actively suicidal
* terminally ill or have
* Dementia
* cognitive impairment
* learning difficulties, or
* the primary care physician knows of another reason to exclude.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Differential contribution of mindfulness for stress and mindfulness for pain courses on Acceptance and Commitment Therapy (ACT) process 1: Acceptance utilising The 7-item Acceptance and Action Questionnaire v.2 | baseline at recruitment; baseline, pre-intervention; during intervention (half-way); immediately after intervention; 3 months after the intervention
  This will be utilised to measure and track the patient's change (if any) - at relevant time points in the study - in willingness to experience general unpleasant feelings and emotions that are not pain related (not to unfairly disadvantage the stress version of the course). Assessed by Likert scale on multiple itemts (1 = Never True ; 7 = Always true)
Differential contribution of mindfulness for stress and mindfulness for pain courses on Acceptance and Commitment Therapy (ACT) process 1a: Pain Acceptance utilisikng the 8-item Chronic Pain Acceptance Questionnaire | baseline, pre-intervention, during intervention, immediately after intervention, 3 months after the intervention
  This will be utilised to measure and track the patient's changes (if any) - at relevant at each time point in the study - with acceptance of pain. Assessed by Likert Scale on multiple items (0 = Never true; 6 = always true).
Differential contribution of mindfulness for stress and mindfulness for pain courses on Acceptance and Commitment Therapy (ACT) process 2: Contact with the Present Moment: The Mindful Attention Awareness Scale will be utilised. | baseline at recruitment; baseline, pre-intervention; during intervention (half-way); immediately after intervention; 3 months after the intervention
  This will be utilised to track and measure the patient's changes (if any) - at each time point in the study - of mindful attention and awareness. Assessed by Liker Scale on multiple items (1 = Almost Always; 6 = Almost Never)
Differential contribution of mindfulness for stress and mindfulness for pain courses on Acceptance and Commitment Therapy (ACT) process 3: Self in context: The Self Experience Questionnaire will be utlised. | baseline at recruitment; baseline, pre-intervention; during intervention (half-way); immediately after intervention; 3 months after the intervention
  This measure will be utilised to track and measure the changes (if any) - at each time point in the study - of patient's ability to observe themselves as separate from triggering processes. Assessed by Likert Scale on multiple items (0 = never true; 6 = always true)
Differential contribution of mindfulness for stress and mindfulness for pain courses on Acceptance and Commitment Therapy (ACT) process 4: Cognitive fusion: the Cognitive Fusion Questionnaire | baseline at recruitment; baseline, pre-intervention; during intervention (half-way); immediately after intervention; 3 months after the intervention
  This will be utilised to measure and track the patient's changes (if any) - at each time point in the study - with how entangled they are with thinking.Assessed by Likert Scale on multiple items (1 = Never True; 7 = always true)
Differential contribution of mindfulness for stress and mindfulness for pain courses on Acceptance and Commitment Therapy (ACT) process 5: Values: The Chronic Pain Values Inventory | baseline, pre-intervention, during intervention, immediately after intervention, 3 months after the intervention
  This will be utilised to measure and track the patient's changes (if any) - at each time point in the study - with how able they are to notice what matters in their life and their discrepancy with / from it. Assessed via Likert scale on importance/success 0 - 5 (0 = not at all important/successful; 5 = extremely important/successful)
Differential contribution of mindfulness for stress and mindfulness for pain courses on Acceptance and Commitment Therapy (ACT) process 6: Committed Action: The 8-item Committed Action Questionnaire | baseline at recruitment; baseline, pre-intervention; during intervention (half-way); immediately after intervention; 3 months after the intervention
  This will be utilised to measure and track the patient's changes (if any) - at each time point in the study - their ability to commit to valuable behaviours. Assessed by likert scale on multiple items (0 = Never True; 6 = always true)

SECONDARY OUTCOMES:
IMMPACT consistent, changes in Pain Intensity (How sore the participant is) will be evaluated utilising the Brief Pain Inventory - Short Form (BPI) | baseline at recruitment; baseline, pre-intervention; during intervention (half-way, week 4 of 8); immediately after intervention; 3 months after the intervention
  1. Pain related distress: The Pain Catastrophizing Scale (Sullivan, Bishop et al. 1995)
  2. Depression: The Beck Depression Inventory - Fast Screen (Poole, Bramwell et al. 2009) Global Impression of Functioning: the Patient's Global Impression of Change (Guy 1976)will allow to consider perceived improvement and deterioration.
  numeric rating scale (NRS) on intensity (scale 0-10) including, worst, least average (in the past week) and right now.
IMMPACT consistent, changes in Pain Interference (on functioning and aspects of quality of life) will be evaluated utilising the Brief Pain Inventory - Short Form (BPI) | baseline at recruitment; baseline, pre-intervention; during intervention (half-way, week 4 of 8); immediately after intervention; 3 months after the intervention
  Numeric rating scale (NRS) on intensity (scale 0-10) including, general activity, mood, ability to get around, normal work, relations with other people, sleep and enjoyment of life. Due to questionnaire burden, the initially planned RMDQ-A and SF-36 will not be administered
IMMPACT consistent measurement of change in emotional functioning: depression screening utilizing the Beck Depression Inventory - Fast Screen (BDI-FS) | baseline at recruitment; baseline, pre-intervention; during intervention (half-way, week 4 of 8); immediately after intervention; 3 months after the intervention
  self-report questionnaire (statements weighted with scores 0 - 3; scores > 5 suggestive of depression)
IMMPACT consistent measurement of change in emotional functioning: catastrophizing, utilizing Pain Catastrophizing Scale (PCS) | baseline at recruitment; baseline, pre-intervention; during intervention (half-way, week 4 of 8); immediately after intervention; 3 months after the intervention
  self-report questionnaire with statements on a Likert Scale; 0 = 'not at all' - 4 = 'all the time').
IMMPACT consistent measurement of change in patient's ratings of global functioning | baseline at recruitment; baseline, pre-intervention; during intervention (half-way, week 4 of 8); immediately after intervention; 3 months after the intervention
  self report questionnaire , utilizing The Patient Global Impressions of Change Scale (PGIC), based on statements scored from 1 = Very Much helped - 7 = Very much worse.
IMMPACT consistent measurement of change in participants' disposition via subjective impression of change on pain, interference from pain, resilience on a scale of -100% (worse) to + 100% better. | baseline at recruitment; baseline, pre-intervention; during intervention (half-way, week 4 of 8); immediately after intervention; 3 months after the intervention
  subjectively reported dispositional changes
IMMPACT consistent measurement of change in pain medication changes utilizing name and amount (mg/g) of pain / mood medication | baseline at recruitment; baseline, pre-intervention; during intervention (half-way, week 4 of 8); immediately after intervention; 3 months after the intervention
  utilising patient reports
Accident and Emergency (A&E) and primary care GP visits | baseline at recruitment; baseline, pre-intervention; during intervention (half-way, week 4 of 8); immediately after intervention; 3 months after the intervention
  patient reported changes in number of GP and hospital visits relating to pain since previously recorded contact as part of the study

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Agostinis, Principal Investigator — Government of Jersey
Locations (1):
- Pain Clinic, Saint Helier, Jersey

REFERENCES:
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Bawa FL, Mercer SW, Atherton RJ, Clague F, Keen A, Scott NW, Bond CM. Does mindfulness improve outcomes in patients with chronic pain? Systematic review and meta-analysis. Br J Gen Pract. 2015 Jun;65(635):e387-400. doi: 10.3399/bjgp15X685297. PMID 26009534
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Abdulla A, Adams N, Bone M, Elliott AM, Gaffin J, Jones D, Knaggs R, Martin D, Sampson L, Schofield P; British Geriatric Society. Guidance on the management of pain in older people. Age Ageing. 2013 Mar;42 Suppl 1:i1-57. doi: 10.1093/ageing/afs200. PMID 23420266
- [Background] Braun V. and Clarke V. (2006) Using thematic analysis in psychology. Qualitative research in Psychology; 3(2):77-101.
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Burch, V. (2008). Living Well with Pain and Illness: Piatkus.
- [Background] Burch, V., & Penman, D. (2013). Mindfulness for Health: A practical guide to relieving pain, reducing stress and restoring wellbeing: Little, Brown Book Group.
- [Background] Day, M. A. (2017). Overview of the eight-session treatment. In Mindfulness-Based Cognitive Therapy for Chronic Pain: A Clinical Manual and Guide, (pp. 89-113): John Wiley & Sons Ltd.
- [Background] Day MA, Jensen MP, Ehde DM, Thorn BE. Toward a theoretical model for mindfulness-based pain management. J Pain. 2014 Jul;15(7):691-703. doi: 10.1016/j.jpain.2014.03.003. PMID 24985483
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Feliu-Soler A, Montesinos F, Gutierrez-Martinez O, Scott W, McCracken LM, Luciano JV. Current status of acceptance and commitment therapy for chronic pain: a narrative review. J Pain Res. 2018 Oct 2;11:2145-2159. doi: 10.2147/JPR.S144631. eCollection 2018. PMID 30323649
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Guyatt GH, Oxman AD, Vist GE, Kunz R, Falck-Ytter Y, Alonso-Coello P, Schunemann HJ; GRADE Working Group. GRADE: an emerging consensus on rating quality of evidence and strength of recommendations. BMJ. 2008 Apr 26;336(7650):924-6. doi: 10.1136/bmj.39489.470347.AD. PMID 18436948
- [Background] Guy W. ECDEU assessment manual for psychopharmacology (DHEW Publication No. ADM 76-338). Washington, DC: US Government Printing Office; 1976.
- [Background] Harrison AM, Scott W, Johns LC, Morris EMJ, McCracken LM. Are We Speaking the Same Language? Finding Theoretical Coherence and Precision in "Mindfulness-Based Mechanisms" in Chronic Pain. Pain Med. 2017 Nov 1;18(11):2138-2151. doi: 10.1093/pm/pnw310. PMID 28082525
- [Background] Hayes SC, Strosahl K, Wilson KG (1999): Acceptance & Commitment therapy: An Experiential Approach to Behaviour Change. New Your, Guilford Press.
- [Background] Hedges, L. (1981). Distribution Theory for Glass's Estimator of Effect Size and Related Estimators. Journal of Educational Statistics, 6(2), 107-128.
- [Background] Hennessy, G. (2017). The Little Mindfulness Workbook: Everyday techniques to help you combat stress and enhance your life: Crimson Publishing.
- [Background] Hilton L, Hempel S, Ewing BA, Apaydin E, Xenakis L, Newberry S, Colaiaco B, Maher AR, Shanman RM, Sorbero ME, Maglione MA. Mindfulness Meditation for Chronic Pain: Systematic Review and Meta-analysis. Ann Behav Med. 2017 Apr;51(2):199-213. doi: 10.1007/s12160-016-9844-2. PMID 27658913
- [Background] Hopper MJ, Curtis S, Hodge S, Simm R. A qualitative study exploring the effects of attending a community pain service choir on wellbeing in people who experience chronic pain. Br J Pain. 2016 Aug;10(3):124-34. doi: 10.1177/2049463716638368. Epub 2016 Mar 22. PMID 27583139
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Kabat-Zinn, J. (2011). Some reflections on the origins of MBSR, skillful means, and the trouble with maps. Contemporary Buddhism, 12(1), 281-306. doi:10.1080/14639947.2011.564844
- [Background] Kabat-Zinn J. Too Early to Tell: The Potential Impact and Challenges-Ethical and Otherwise-Inherent in the Mainstreaming of Dharma in an Increasingly Dystopian World. Mindfulness (N Y). 2017;8(5):1125-1135. doi: 10.1007/s12671-017-0758-2. Epub 2017 Jun 29. No abstract available. PMID 28989546
- [Background] MBSR Course Outline. (2017). Retrieved from https://www.umassmed.edu/cfm/mindfulness-based-programs/mbsr-courses/mbsr/mbsr-course-outline/
- [Background] MBTT. (2011). Good Practice Guidelines for Teaching Mindfulness Based Courses. In: UK Network for Mindfulness Based Teachers.
- [Background] McCracken LM, Sato A, Taylor GJ. A trial of a brief group-based form of acceptance and commitment therapy (ACT) for chronic pain in general practice: pilot outcome and process results. J Pain. 2013 Nov;14(11):1398-406. doi: 10.1016/j.jpain.2013.06.011. Epub 2013 Sep 12. PMID 24035351
- [Background] McCracken LM, Vowles KE. Acceptance and commitment therapy and mindfulness for chronic pain: model, process, and progress. Am Psychol. 2014 Feb-Mar;69(2):178-87. doi: 10.1037/a0035623. PMID 24547803
- [Background] Morse, J. M. (2000). Determining Sample Size. Qualitative Health Research, 10(1), 3-5.
- [Background] Nicholas MK. Self-efficacy and chronic pain. In Paper presented at the annual conference of the British Psychological Society, St. Andrews, Scotland; 1989.
- [Background] Poole H, Bramwell R, Murphy P. The utility of the Beck Depression Inventory Fast Screen (BDI-FS) in a pain clinic population. Eur J Pain. 2009 Sep;13(8):865-9. doi: 10.1016/j.ejpain.2008.09.017. Epub 2008 Nov 14. PMID 19010075
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Santorelli, S., F. (2014). Mindfulness-Based Stress Reduction (MBSR): Standards of Practice. In. Division of Preventive and Behavioral Medicine, University of Massachussets Medical School: The Centre for Mindfulness, Medicine, Health Care and Society.
- [Background] Scott W, McCracken LM, Norton S. A Confirmatory Factor Analysis of Facets of Psychological Flexibility in a Sample of People Seeking Treatment for Chronic Pain. Ann Behav Med. 2016 Apr;50(2):285-96. doi: 10.1007/s12160-015-9752-x. PMID 26608280
- [Background] Segal, Z., V., Williams, J. M. G., & Teasdale, J., D. (2002). Mindfulness-based cognitive therapy for depression: A new approach to preventing relapse. New York, NY, US: Guilford Press.
- [Background] Shapiro SL, Carlson LE, Astin JA, Freedman B. Mechanisms of mindfulness. J Clin Psychol. 2006 Mar;62(3):373-86. doi: 10.1002/jclp.20237. PMID 16385481
- [Background] Sullivan, M.J.L., Bishop, S. and Pivik, J. (1995) The Pain Catastrophizing Scale: Development and Validation. Psychological Assessment, 7, 524-532.
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Van Dam NT, van Vugt MK, Vago DR, Schmalzl L, Saron CD, Olendzki A, Meissner T, Lazar SW, Kerr CE, Gorchov J, Fox KCR, Field BA, Britton WB, Brefczynski-Lewis JA, Meyer DE. Mind the Hype: A Critical Evaluation and Prescriptive Agenda for Research on Mindfulness and Meditation. Perspect Psychol Sci. 2018 Jan;13(1):36-61. doi: 10.1177/1745691617709589. Epub 2017 Oct 10. PMID 29016274
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Yu, L., McCracken, L. M., & Norton, S. (2016). The Self Experiences Questionnaire (SEQ): Preliminary analyses for a measure of self in people with chronic pain. Journal of Contextual Behavioral Science, 5(3), 127-133. doi:10.1016/j.jcbs.2016.07.006
- [Background] Kabat-Zinn, J. (2013). Full catastrophe living: using the wisdom of your body and mind to face stress, pain, and illness. Rev. and updated edition, Bantam Books trade paperback edition. New York: Bantam Books.
- [Background] BPS (2013) Guidelines for pain management programmes for adults. British Pain Society. https://www.britishpainsociety.org [Free Full-text]
- [Background] Dobkin PL. Mindfulness-based stress reduction: what processes are at work? Complement Ther Clin Pract. 2008 Feb;14(1):8-16. doi: 10.1016/j.ctcp.2007.09.004. Epub 2007 Nov 13. PMID 18243937
- [Background] Williams L. Mindfulness on pain management programmes - are we teaching it as well as we could? Pain News.2019; 17(1) 31-32
- [Background] Fish RA, McGuire B, Hogan M, Morrison TG, Stewart I. Validation of the chronic pain acceptance questionnaire (CPAQ) in an Internet sample and development and preliminary validation of the CPAQ-8. Pain. 2010 Jun;149(3):435-443. doi: 10.1016/j.pain.2009.12.016. Epub 2010 Feb 25. PMID 20188472
- [Background] McCracken LM, Yang SY. The role of values in a contextual cognitive-behavioral approach to chronic pain. Pain. 2006 Jul;123(1-2):137-45. doi: 10.1016/j.pain.2006.02.021. Epub 2006 Mar 29. PMID 16564627
- [Background] Yu L, Scott W, Goodman R, Driscoll L, McCracken LM. Measuring 'self': preliminary validation of a short form of the Self Experiences Questionnaire in people with chronic pain. Br J Pain. 2021 Nov;15(4):474-485. doi: 10.1177/2049463721994863. Epub 2021 Feb 19. PMID 34840795
- [Background] McCracken LM, Chilcot J, Norton S. Further development in the assessment of psychological flexibility: a shortened Committed Action Questionnaire (CAQ-8). Eur J Pain. 2015 May;19(5):677-85. doi: 10.1002/ejp.589. Epub 2014 Sep 2. PMID 25181605
- [Background] Sullivan, M. J. L., S. R. Bishop and J. Pivik (1995).

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05498454/Prot_SAP_ICF_000.pdf